CLINICAL TRIAL: NCT06761651
Title: TAVO412 a Two-stage, Open-label, Phase I Study in Patients with Advanced/metastatic Solid Tumors Who Have Received Standard of Care
Brief Title: A Study of TAVO412 in Patients with Cancer (TAVO412)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tavotek Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59870005
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Cancer
Keywords: TAVO412
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part 1 Cohort1 (Other): 150mg bi-weekly IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 1 Cohort2 (Other): 375mg bi-weekly IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 1 Cohort3 (Other): 750mg bi-weekly IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 1 Cohort4 (Other): 1125mg bi-weekly IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 1 Cohort5 (Other): 1500mg bi-weekly IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 2 Cohorts (Other): RP2D IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 1 Cohort6 (Other): 1750mg bi-weekly IV infusion of TAVO412
  Interventions: Drug: TAVO412

INTERVENTIONS:
Drug: TAVO412 — Biologic

SUMMARY:
TAVO412 Phase 1 is an open-label, non-randomized, 2-part Phase I study to examine the safety, tolerability, pharmacokinetics/pharmacodynamics, and preliminary efficacy of TAVO412. Part 1 will utilize a standard 3 + 3 design to determine the MTD/RP2D of TAVO412 in subjects with advanced or metastatic solid tumors who progressed on prior approved standard of care therapy. Part 2 will further evaluate the safety, tolerability, preliminary efficacy, pharmacokinetics (PK), and pharmacologic activity of TAVO412 in a new set of subjects with advanced or metastatic gastric cancer, non-small cell lung cancer (NSCLC), or subjects of other solid tumor types with best clinical responses (e.g., CR > PR > SD) from Part 1 that progressed on prior approved standard of care therapy.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, Phase I study to determine the safety and tolerability, define the MTD/RP2D, and assess the preliminary efficacy of TAVO412 in subjects with advanced or metastatic solid tumors who progressed on prior approved standard of care therapy. Subjects will receive TAVO412 at the tested dose intravenously on Day 1 and 15 in Cycle 1 and will continue this bi-weekly treatment schedule for all future cycles.

The study will be conducted in 2 parts:

Part 1 - Dose Escalation will determine the MTD and/or RP2D of TAVO412, which includes defining the optimal dose administration schedule.

Part 2 - Cohort Expansion will evaluate the recommended dose and administration schedule (MTD/RP2D) determined in Part 1 in a new set of subjects with advanced or metastatic gastric cancer, non-small cell lung cancer (NSCLC), or subjects of other solid tumor types with best clinical responses (e.g., CR > PR > SD) from Part 1 that progressed on prior approved standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male/female 18 years of age or older at the time of screening. 2. Voluntarily signed informed consent, understand the study and are willing to follow and have the ability to complete all trial procedures.

  3. Subjects with histologically or cytologically pathologically confirmed locally advanced unresectable or metastatic solid tumors that have failed standard therapy or have no standard therapy. There is no limit to the number of treatments that can be used in a previous regimen.

  4. ECOG performance status 0 or 1. 5. Expected survival ≥ 3 months. 6. Participants enrolled in Phase 2 must have at least one measurable (RECIST v1.1 criteria) lesion, and participants enrolled in Phase 1 may also be enrolled if only non-measurable (RECIST v1.1 criteria) lesions are present. Neoplastic lesions located in the field of prior radiation therapy or treated with other local therapies are not considered measurable unless disease progression has been demonstrated.

  7. Phase 1: Subjects with advanced or metastatic solid tumors who have failed standard therapy or have no standard treatment.

  8. Phase 2: A new cohort of subjects with advanced or metastatic solid tumors who have failed or had no standard therapy and are of high prevalence in China, such as non-small cell lung cancer, gastric cancer, and liver cancer, or other solid tumor types with the best clinical response observed from Phase 1 (e.g., CR > PR > SD).
  1. For subjects with non-small cell lung cancer: histologically or cytologically confirmed non-small cell lung cancer with mutations or gene amplification in EGFR, MET, or VEGF genes, EGFR or cMET overexpression (refer to IHC≥2+ in the Central Laboratory Immunohistochemistry Antibody Interpretation Criteria, ≥ intermediate staining).
  2. For subjects with gastric cancer: histopathologically confirmed gastric cancer or gastroesophageal junction cancer (including lower esophageal adenocarcinoma) with mutations or gene amplifications in EGFR, MET, or VEGF genes, EGFR or cMET overexpression (IHC≥2+ in reference central laboratory immunohistochemistry antibody interpretation criteria, ≥ moderate staining).
  3. For subjects with hepatocellular carcinoma: histologically or cytologically pathologically confirmed primary hepatocellular carcinoma with mutations or gene amplification in EGFR, MET or VEGF, overexpression of EGFR or cMET (IHC≥2+ in reference central laboratory immunohistochemistry antibody interpretation standards, ≥ moderate staining).

Note: The tumor biopsy test report performed by the subject for other purposes (i.e., not a protocol-defined procedure) within 1 year prior to signing the consent form can be used as the basis for pre-treatment biopsy evaluation, and if metastases or recurrences of other tumors have occurred within 1 year, they are excluded.

9. Stage 2: Willing to undergo pre-treatment and end-of-treatment (if appropriate) tumor biopsy (rough needle aspiration or excision) of a tumor tissue sample for biomarker immunohistochemistry and genetic testing.

Note: Tumor biopsy archival tissue samples performed by subjects for other purposes (i.e., not protocol-defined procedures) within 1 year prior to signing the consent form may be used as pre-treatment tumor biopsy tissue samples, excluded if metastases or recurrences of other tumors have occurred within 1 year.

Note: Subjects are required to provide 4-6 blank sections with a layer thickness of 3-5 μm and 10-12 blank sections with a layer thickness of 8-10 μm, or preferably 1 tissue block for EGFR and cMET immunohistochemistry and polygenic mutation/amplification detection. If the amount of tumor tissue obtained is limited, it is important to prioritize the need for EGFR and cMET immunohistochemistry detection (at least 4 blank sections with a layer thickness of 3-5 μm), followed by tumor tissue polygenic detection (10-12 blank sections with a layer thickness of 8-10 μm), and finally FISH detection for EGFR and MET gene amplification of tumor tissue (4-6 blank sections with a thickness of 3-5 μm).

Note: Pre-treatment tumor tissue sections are not mandatory for subjects in Phase 2 if the tumor biopsy test report for other purposes (i.e., not a protocol-defined procedure) within 1 year prior to signing the consent form contains EGFR or cMET immunohistochemistry results. At the end of treatment, it is not suitable for/unwilling to provide tissue samples or other reasons that preclude tumor biopsy, and tumor biopsy is not mandatory.

Note: Tumor tissue samples are optional before and at the end of treatment in Phase 1, and best efforts should be made to obtain tumor tissue if possible. Test results are collected if the subject has had a tumor biopsy for other purposes (i.e., not a protocol-defined procedure) within 1 year prior to signing the consent form, and the test results contain EGFR, cMET, or VEGF.

10. For Phase 1 and Phase 2, subjects agree to collect additional peripheral blood for circulating tumor cell DNA (ctDNA) analysis.

11. Female subjects of childbearing potential (defined as not undergoing hysterectomy and/or bilateral oophorectomy sterilization surgery and not postmenopausal, menopausal is defined as amenorrhea ≥ 12 months) must have a negative blood pregnancy test at screening.

1. All female subjects of childbearing potential must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening until 60 days after the last dose of study drug is administered. Male partners of female subjects (other than men who have been sterilized) must agree to use condoms correctly and on a continuous basis for the duration of the study and for 60 days after receiving the last dose of study drug.
2. All male subjects (except those who have been sterilized) must agree to take appropriate precautions to avoid pregnancy with their partner (with at least 99% certainty) from screening until 90 days after the last dose of study drug administration. The female partner of male subjects (if of childbearing potential or less than 12 months postmenopausal) must agree to use a highly effective method of contraception for the duration of the study and within 90 days of receiving the last dose of study drug. In addition, sperm donation is not allowed during the study and for 90 days after receiving the last dose of study drug.
3. At least 99% effective contraceptive methods (see Appendix A) should be communicated to subjects and their understanding confirmed.

   12. All of the following criteria need to be met during the screening period, and if the following screening laboratory tests were performed > 7 days prior to the start of treatment, they will need to be repeated within 7 days prior to the start of treatment.

a. Absolute neutrophil count ≥ 1.5 ×109/L, platelet ≥ 100 ×109/L, hemoglobin ≥9 g/dL or ≥5.6 mmol/L, and no transfusion of blood products (including platelets or red blood cells) or use of colony-stimulating factors (including granulocyte colony-stimulating factor, Granulocyte macrophage colony-stimulating factor or recombinant erythropoietin) (the washout period of long-acting colony-stimulating factor or erythropoietin is at the discretion of the investigator).

b. AST and ALT≤2.5×Upper limit of normal(ULN)(AST and ALT in subjects with primary or metastatic liver cancer≤5× ULN)。 c. Total bilirubin ≤ 1.5 × ULN (3× ULN for subjects with Gilbert's syndrome ≤), if there is no ULN at the study institution, direct bilirubin must be < 40% of total bilirubin.

d. Creatinine clearance ≥ 30 mL/min (estimated by the Cockcroft-Gault formula, [140-age]× weight (Kg)/serum creatinine (mg/dl) × 72, or [140-age]× body weight (Kg)/serum creatinine (μmol/L) × 0.818, calculated × 0.85 for women).

e. International normalized ratio (INR) ≤ 1.5× ULN, activated partial thromboplastin time (APTT) ≤ 1.5×ULN (without anticoagulant); INR ≤2.5×ULN, APTT≤2.5×ULN (those using anticoagulants).

13. Human immunodeficiency virus (HIV)/hepatitis B (HBV)/hepatitis C (HCV) subjects will be allowed to participate in the study if the following criteria are met:

1. HIV-infected subjects: CD4+ T cell (CD4+) count must be ≥ 350 cells/μL; Subjects with HIV infection-related tumors (e.g., Kaposi's sarcoma and invasive cervical cancer) were allowed to enroll; To ensure that subjects can tolerate effective antiretroviral therapy and that toxicity is not confused with study drug toxicity, subjects should receive at least four weeks of established antiretroviral therapy prior to enrollment and have an HIV viral load of less than 400 copies/mL and require replacement of specific ART drugs that may have overlapping toxicity or interaction with the study drug, and exclusion if no replaceable drug is available.
2. Subjects who have no history of hepatitis B infection but have been vaccinated against hepatitis B and have tested positive for hepatitis B surface antibody by serology can participate in the study; HBV virus carriers or subjects with chronic active hepatitis B, whose HBV-DNA copy number is lower than the lower limit of normal in each center after anti-hepatitis B virus treatment, and whose liver function meets the above requirements can participate in the study.
3. If the subject is positive for hepatitis C antibody, the HCV-RNA is lower than the lower limit of normal after drug treatment, and the subject is not at risk of hepatic insufficiency, he or she can participate in the study.

   Note: Viral replication and possible interactions and overlapping toxicities of antiviral therapy with the study drug should be closely monitored during the study participation in the above three categories of subjects

   Exclusion Criteria:
   * 1. Prior to the first dose of study drug, received an anticancer drug or investigational drug at the following time intervals:

     * Chemotherapy, targeted small molecule therapy, or radiotherapy ≤ 14 days. Subject requires long-term corticosteroid use and develops radiation pneumonitis as a result of radiotherapy. A washout period of 1 week after palliative radiotherapy for non-central nervous system (CNS) disease is allowed with the approval of the sponsor. Note: The investigator can judge the washout period at the discretion of the subject according to the subject's condition and the nature of the drug; TKI drugs have a short half-life, and the washout period is more than 5 half-lives.

   Note: Bisphosphonates and denosumab are allowed concomitant medications. • ≤ immunotherapy or cell therapy prior to 28 days (i.e., chimeric antigen receptor T cell therapy; Other cell therapies must be discussed with the investigator to determine eligibility).
   * ≤ Monoclonal antibodies used for anticancer therapy prior to 28 days, with the exception of denosumab.
   * ≤ Chinese medicine used for anti-tumor before 14 days.
   * ≤ 7 days for immunosuppressive therapy for any reason. Note: The use of inhaled or topical steroids or corticosteroids for imaging procedures is permitted.

   Note: Physiologic corticosteroid replacement therapy may be approved after consultation with the investigator (systemic prednisone or equivalent corticosteroid doses of ≤10mg/day are allowed).

   • All other investigational drugs or devices are ≤ 28 days or 5 half-lives (whichever is longer) prior to the first dose. For investigational drugs with longer half-lives (e.g., > 5 days), investigator approval is required for enrollment prior to the fifth half-life.

   2. Have not recovered from the toxic effects of prior therapy (including prior immunotherapy) and/or complications of surgical intervention to CTCAE v5.0 score ≤ Grade 1.

   Note: Subjects with stable chronic AEs (≤ Grade 2) that are not expected to resolve spontaneously (e.g., peripheral neuropathy and alopecia) are exceptions and may be enrolled after receiving investigator approval.

   Note: Subjects with a history of clinically symptomatic ocular disease judged by the investigator to be severe or uncontrollable will be excluded, including but not limited to severe or uncontrollable keratitis, dry eye syndrome, conjunctivitis, blurred vision, visual impairment, uveitis, etc.

   Note: Subjects with a history of prior therapy-related Grade 3 or higher AEs (excluding hematologic AEs) are excluded from the dose escalation portion of the study. The investigator can analyze the AE according to the time of occurrence and recovery.

   3. Other malignant tumors at the same time, such as tumors that occurred and cured 5 years ago, do not affect enrollment: melanoma, skin cancer, carcinoma in situ or non-invasive tumors.

   4. Previous clinically significant cardiac disease within 6 months prior to the first study drug administration, including:
   * i. myocardial infarction, ii. Unstable angina, iii. Cerebrovascular accident, iv. Other acute uncontrollable cardiac disease;
   * History of clinically significant ventricular arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes);
   * New York Heart Association (NYHA) Class III or IV congestive heart failure;
   * QTcF ≥470ms (Female) or≥450ms (Male) Or congenital long QT syndrome history or family history（Naring A，2012）；
   * Arrhythmias requiring anti-arrhythmic drug therapy (subjects with atrial fibrillation with controlled heart rate > 1 month prior to the first dose of trial drug are eligible for enrollment); 5. Subjects who require local treatment or repeated drainage, and who are judged by the investigator to have poorly controlled effusions in body cavities (pleural effusion, ascites, pericardial effusion, etc.).

     6. Patients with recent gastrointestinal bleeding (defined as a history of hematemesis, visible hematochezia, or melena within the past 3 months (including hematochezia or melena due to hemorrhoids) without evidence of recovery confirmed by endoscopy or colonoscopy).

     7. Those with evidence of gastric bleeding or gastric perforation who will be excluded from participation at the discretion of the investigator.

     8. Those with pyloric obstruction or persistent recurrent vomiting (defined as vomiting ≥ 3 times in 24 hours) or those with acute intestinal obstruction are intubated.

     9. Those with a previous history of ulcerative colitis or Crohn's disease. 10. Those who have had active colitis, including infectious colitis, radiation colitis, and ischemic colitis, within 4 weeks prior to screening.

     11. Received a live vaccine within 30 days of the start of the study drug program.

   Note: Types of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/shingles, yellow fever, rabies, BCG, and typhoid vaccines. Seasonal influenza vaccines for injection are generally inactivated vaccines and are allowed; COVID-19 booster vaccine ≥ 4 weeks after the end of the study is allowed; However, intranasal influenza vaccine is a live-attenuated vaccine and is not allowed.

   12. Active autoimmune disease requiring systemic therapy (i.e., use of immunomodulators, corticosteroids, or immunosuppressive medications).

   Note: Subjects who have not required systemic therapy in the past 2 years should discuss their condition with the investigator to determine enrollment.

   Note: Subjects with hyperthyroidism/hypothyroidism may participate. Note: Hormone replacement therapy and symptomatic therapy (e.g., levothyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are not considered a form of systemic therapy and are permitted.

   13. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

   Note: Subjects with previously treated brain metastases may participate provided that they are stable (no evidence of radiographic progression for at least 28 days prior to the first dose of study drug, and any neurological symptoms have returned to normal values), no evidence of new or enlarging brain metastases or central nervous system edema, and no steroid therapy or antiepileptic therapy is required for at least 14 days prior to the first dose of study drug.

   14. Evidence of active non-infectious pneumonitis or interstitial pneumonitis during the screening period. Subjects who have suffered from interstitial pneumonia in the past and have recovered after treatment can be enrolled in this study after evaluation by the investigator.

   15. Known serious vascular embolic event requiring medical or surgical intervention (≥ grade 2).

   16. Active infection requiring systemic treatment, including COVID-19. 17. Known allergic reaction to any component of the study drug or formulation. 18. Females who are pregnant or lactating, or who are expected to become pregnant from the start of the screening visit until 60 days after the last 1 dose of study drug; 19. Men who plan to impregnate their partner from the start of the screening visit until 90 days after the last dose of study drug.

   20. Any condition that, in the judgment of the investigator, would interfere with full participation in the study, including the use of study drugs and participation in required study visits; poses a significant risk to the subject; or interfere with the interpretation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of TAVO412 according to Adverse Events and Number of Participants With Dose Limiting Toxicity (DLT) using National Cancer Institute CTCAE v5.0 | Approximately 12 months
  According to the frequency, duration, and severity of Adverse Events (AEs). The Dose Limiting Toxicity (DLT) is based on drug related adverse events and includes unacceptable hematologic toxicity, non-hematologic toxicity of Grade 3 or higher, or elevations in hepatic enzymes suggestive of drug-induced liver injury.
  The Common Terminology Criteria for Adverse Events (CTCAE) v5.0 has a minimum value of Grade 1, or mild, and a maximum value of Grade 4, Life-threatening; pressor or ventilatory support indicated. All DLTs will be assessed by the investigator using National Cancer Institute CTCAE v5.0.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of TAVO412 | Approximately 12 months
  The Cmax is the maximum observed serum concentration of TAVO412.
Time to Reach Maximum Observed Serum Concentration (Tmax) of TAVO412 | Approximately 12 months
  The Tmax is defined as time to reach maximum observed serum concentration of TAVO412.
Minimum Serum Concentration (Cmin) of TAVO412 | Approximately 12 months
  The Cmin is the minimum observed serum concentration of TAVO412.
Area Under the Serum Concentration-Time Curve From 0-1 (AUC[t0-t1]) | Approximately 12 months
  The AUC(t0-t1) is the area under the serum TAVO412 concentration-time curve from time t0 to t1.
Overall Response Rate (ORR) | Approximately 12 months
  Overall Response Rate (ORR)
Duration of Response (DOR) | Approximately 12 months
  DOR is defined as the time from earliest date of disease response (CR or PR) until earliest date of disease progression.
Progression-Free Survival (PFS) | Approximately 12 months
  PFS is defined as the time from date of first dose of study drug until the earliest date of disease progression.
Duration of Disease Control (CR, PR, and SD) | Approximately 12 months
  Duration of disease control is defined as the sum of PFS followed by maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Dr., Principal Investigator — Henan Cancer Hospital
Locations (6):
- China (6):
  - Affiliated Cancer Hospital of Chongqing University, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Jinan Central Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No
Legal restriction